CLINICAL TRIAL: NCT00638989
Title: An Open-Label, Parallel-Group, Bioavailability Study to Assess the Pharmacokinetics of CAT-354 Following Subcutaneous and Intravenous Administration
Brief Title: A Study to Assess Bioavailability and Pharmacokinetics of CAT- 354
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAT-354-0703
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Asthma; Healthy
Keywords: Asthma; CAT-354; Tralokinumab; Healthy
MeSH Terms: conditions — Asthma | interventions — tralokinumab; Injections, Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CAT-354 150 mg (intravenous) (Experimental): A single dose of CAT-354 150 milligram (mg) intravenous infusion over 30 minutes on Day 0.
  Interventions: Biological: CAT-354 150 mg (intravenous)
- CAT-354 150 mg (subcutaneous) (Experimental): A single dose of CAT-354 150 mg injection subcutaneously on Day 0.
  Interventions: Biological: CAT-354 150 mg (subcutaneous)
- CAT-354 300 mg (subcutaneous) (Experimental): A single dose of CAT-354 300 mg injection subcutaneously on Day 0.
  Interventions: Biological: CAT-354 300 mg (subcutaneous)

INTERVENTIONS:
Biological: CAT-354 150 mg (intravenous) — A single dose of CAT-354 150 milligram (mg) intravenous infusion over 30 minutes on Day 0.
  Other Names: Tralokinumab
  Arms: CAT-354 150 mg (intravenous)
Biological: CAT-354 150 mg (subcutaneous) — A single dose of CAT-354 150 mg injection subcutaneously on Day 0.
  Other Names: Tralokinumab
  Arms: CAT-354 150 mg (subcutaneous)
Biological: CAT-354 300 mg (subcutaneous) — A single dose of CAT-354 300 mg injection subcutaneously on Day 0.
  Other Names: Tralokinumab
  Arms: CAT-354 300 mg (subcutaneous)

SUMMARY:
To compare bioavailability and pharmacokinetics of CAT-354 following subcutaneous administration compared with intravenous administration.

DETAILED DESCRIPTION:
To compare the bioavailability and pharmacokinetics of CAT-354 following subcutaneous administration of 150 milligram (mg) and 300 mg compared with 150 mg given intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent is obtained prior to any study related procedure taking place
* Males, aged 19-55 years
* No significant abnormality on clinical examination or medical history (excluding atopic skin signs, symptoms and history)
* A normal 12-lead electrocardiogram (ECG) (no clinically significant abnormalities)
* Clinical chemistry, hematology and urinalysis results within the laboratory reference ranges or deemed not clinically significant by the Investigator
* A negative screen for drugs of abuse and alcohol
* Body mass index (BMI) between 18-30 kilogram per square meter (kg/m^2), inclusive
* No other clinically significant abnormality on history and clinical examination
* Able to comply with the requirements of the protocol.

Exclusion Criteria:

* Any active concomitant disease including psychological disorders
* History of medication that might carry over effects into study
* Previously received monoclonal antibody, or a similar related protein, that might sensitize subjects to CAT-354
* Participation in another investigational medicinal product study within 3 months of the start of this study or 5 half-lives of the previously administered investigational medicinal product (IMP), whichever is the longer except methodological studies in which no IMP was given
* Any acute illness in the 2 weeks before Day 0 (Visit 2)
* Any blood donation or significant loss of blood within 56 days of study initiation or plasma donation within 7 days of study initiation
* Subject is a participating Investigator, sub-Investigator, study coordinator, or employee of a participating Investigator, or is a first degree relative of the aforementioned
* Any factor which, in the opinion of the Investigator, would jeopardize the evaluation or safety or be associated with poor adherence to the protocol
* The subject's primary care physician recommends the subject should not take part in the study
* Subjects with immunodeficiency disorders
* Subjects who have a positive test for, or have been treated for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04-11 (Actual); Primary Completion 2008-06-07 (Actual); Study Completion 2008-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (1):
- MDS Pharma Services (US) Inc., Lincoln, Nebraska, United States

REFERENCES:
- [Background] Oh CK, Faggioni R, Jin F, Roskos LK, Wang B, Birrell C, Wilson R, Molfino NA. An open-label, single-dose bioavailability study of the pharmacokinetics of CAT-354 after subcutaneous and intravenous administration in healthy males. Br J Clin Pharmacol. 2010 Jun;69(6):645-55. doi: 10.1111/j.1365-2125.2010.03647.x. PMID 20565456

RESULTS

PARTICIPANT FLOW:
Groups:
- CAT-354 150 mg (Subcutaneous): A single dose of CAT-354 150 mg injection, subcutaneously on Day 0.
Period: Overall Study
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Started | 10 | 10 | 10
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous) | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (8.3) | 39.3 (8.6) | 27.8 (10.4) | 32.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability of CAT-354 After Subcutaneous Dose
Description: Bioavailability (F) is a measurement of the rate and extent to which a drug reaches the systemic circulation. Absolute bioavailability of the subcutaneous doses was assessed by the geometric least-square means ratios of subcutaneous to intravenous dose-normalized area under the serum concentration-time curve from time zero to infinity (AUC [0 - infinity]/Dose). AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: Predose, end of infusion, 30 minutes, 1, 3, 8 and 24 hours post-end of infusion/post-injection on Day 0; Day 3, 5, 7, 9, 14, 21, 28, 35, 42 and 56
Population: Pharmacokinetic (PK) population included all evaluable participants who received at least 1 dose of study medication and had sufficient post-dose blood samples to estimate maximum observed serum concentration (Cmax).
Measure: Geometric Mean (90% Confidence Interval); unit: percent bioavailability
Arm/Group | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10
percent bioavailability | 62.1 [48.5 to 79.6] | 60.1 [46.9 to 77.1]

2. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and up to Day 56 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 0 to 56
Population: Safety population included all participants randomized to treatment, and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
participants
  TEAEs | 5 | 5 | 4
  TESAEs | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies for CAT-354 at Any Visit
Time Frame: Day 0 and Day 56
Population: Safety population included all participants randomized to treatment, and received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
participants | 0 | 0 | 0

4. Secondary Outcome: Area Under the Concentration-time Curve From Zero to Infinity (AUC [0 - Infinity])
Description: AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity).
Time Frame: as for outcome 1
Population: PK population included all evaluable participants who received at least 1 dose of study medication and had sufficient post-dose blood samples to estimate Cmax.
Measure: Mean (Standard Deviation); unit: (microgram*day)/milliliter (mcg*day/mL)
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
(microgram*day)/milliliter (mcg*day/mL) | 903 (291) | 548 (143) | 1080 (315)

5. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC[0 - 56])
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
mcg*day/mL | 765 (220) | 467 (122) | 881 (287)

6. Secondary Outcome: Dose Normalized Area Under the Concentration-time Curve From Zero to Infinity ([AUC {0 - Infinity}]/Dose)
Description: AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity). (AUC [0 - infinity]) was normalized by CAT-354 dose.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ([mcg*day]/mL)/mg
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
([mcg*day]/mL)/mg | 6.02 (1.94) | 3.66 (0.953) | 3.59 (1.05)

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
microgram/milliliter (mcg/mL) | 58.3 (14.4) | 17.1 (5.91) | 36.6 (13.1)

8. Secondary Outcome: Dose Normalized Maximum Observed Concentration (Cmax/Dose)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: (mcg/mL)/mg
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
(mcg/mL)/mg | 0.389 (0.096) | 0.114 (0.039) | 0.122 (0.044)

9. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
days | 0.063 [0.042 to 1.02] | 5 [3 to 9] | 5 [3 to 9]

10. Secondary Outcome: Terminal Phase Elimination Half Life (t1/2)
Description: Terminal phase elimination half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10 | 10
days | 21.4 (2.46) | 19.2 (3.1) | 19.4 (3.59)

11. Secondary Outcome: Apparent Systemic Clearance (CL/F) After Subcutaneous Dose
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after subcutaneous dose (apparent systemic clearance) is influenced by the fraction of the dose absorbed (bioavailability).
Time Frame: Predose, 30 minutes, at 1, 3, 8 and 24 hours post-injection on Day 0; Day 3, 5, 7, 9, 14, 21, 28, 35, 42 and 56
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Number analyzed (Participants) | 10 | 10
mL/day | 292 (82.3) | 307 (109)

12. Secondary Outcome: Apparent Systemic Clearance (CL/F) After Intravenous Dose
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Predose, end of infusion, 30 minutes, 1, 3, 8 and 24 hours post-end of infusion on Day 0; Day 3, 5, 7, 9, 14, 21, 28, 35, 42 and 56
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | CAT-354 150 mg (Intravenous)
Number analyzed (Participants) | 10
mL/day | 188 (84.0)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) After Intravenous Infusion
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Volume of distribution at steady state (Vss) after intravenous dosing was estimated by the formula Vss=MRT(Infinity)*CL, where MRT(Infinity)= AUCM(Infinity)/AUC(0 - infinity) where MRT(Infinity) = mean residence time at infinity, CL= clearance, AUCM[Infinity] = area under the moment curve, and AUC (0 - infinity) = area under the serum concentration versus time curve from time zero (predose) to extrapolated infinite time (0 - infinity).
Time Frame: Predose, end of infusion, 30 minutes, at 1, 3, 8 and 24 hours post-end of infusion on Day 0; Day 3, 5, 7, 9, 14, 21, 28, 35, 42 and 56
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CAT-354 150 mg (Intravenous)
Number analyzed (Participants) | 10
mL | 4960 (1440)

ADVERSE EVENTS:
Time Frame: Day 0 to 56
Arm/Group | CAT-354 150 mg (Intravenous) | CAT-354 150 mg (Subcutaneous) | CAT-354 300 mg (Subcutaneous)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 5/10 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAT-354 150 mg (Intravenous) (N=10) | CAT-354 150 mg (Subcutaneous) (N=10) | CAT-354 300 mg (Subcutaneous) (N=10)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 4 (7) | 1 (3)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hype (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pharyngolaryngeal pa (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.